CLINICAL TRIAL: NCT02046590
Title: A Randomized Controlled Trial (RCT) of Efficacy and Safety of Sedation Compared to General Anesthesia for Endoscopic Retrograde Cholangio-pancreatography
Brief Title: RCT of Efficacy and Safety of Sedation Compared to General Anesthesia for ERCP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too slow
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, vincent huberty, MD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B406201318623
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia; ERCP; Safety; Efficacy
Keywords: Propofol; remifentanil; safety; gastro-intestinal; ERCP; minimally invasive; intubation; ventilation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Propofol; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep Sedation (Active Comparator): Remifentanil 1ng/ml throughout the procedure. Propofol administration starts at an initial (estimated plasma) target concentration of 1,5 microg/ml.
  Propofol administration is adjusted to level 1 or 2 on the modified observer's assessment of alertness/sedation scale. The propofol infusion will be increased stepwise by 0,5 microg/ml every 1 minute until loss of consciousness. Propofol is continued while maintaining spontaneous ventilation without assistance and systolic blood pressure ≥ 60 % of baseline systolic blood pressure.
  Interventions: Drug: Propofol
- General Anaesthesia (Active Comparator): General anesthesia will be induced with target controlled infusion (TCI) of propofol and remifentanil as in the group "deep sedation".
  Suxamethonium (succinylcholine) will be used to facilitate intubation. Endotracheal tube balloon pressure will be controlled during the procedure. Ventilation will be assisted using 40% oxygen in air mixture and mechanically controlled using an anaesthetic ventilator.
  Interventions: Other: General anesthesia

INTERVENTIONS:
Drug: Propofol
  Arms: Deep Sedation
Other: General anesthesia
  Arms: General Anaesthesia

SUMMARY:
There is a worldwide trend to minimally invasive interventions, which results in increasing numbers of interventions performed outside of the operating room. Currently, approximately 12 to 15% of total anaesthetic workload is non-operating room anaesthesia (NORA) and this anaesthetic activity is increasing.

Many of these interventions need supplementary comfort measures to have relaxed patients and high success rates. Endoscopic retrograde cholangio-pancreatography (ERCP) is performed >50,000 times per year in the U.S.,and is a typical minimally invasive intervention that needs patient sedation.

There is a controversy about the optimal comfort intervention in minimally invasive interventions and in particular in ERCP. Two different approaches to insure patients' comfort have been proposed: general anaesthesia with endotracheal intubation and mechanical ventilation or sedation with spontaneous ventilation.

Well-performed studies on sedation versus general anaesthesia using a randomized controlled trial design with observer blinding will contribute to improve the decision-making for the optimal comfort measures in minimally invasive procedures. At our knowledge such a randomized controlled trial has not been reported before. The investigators hypothesize that deep sedation without tracheal intubation will achieve similar success rates for ERCP as general anaesthesia and will have similar rates of harmful postoperative effects.

The primary aim of this trial is to demonstrate that the success rate of ERCP is not inferior in patients randomized to deep sedation without orotracheal intubation vs general anesthesia with orotracheal intubation. Secondary aims include a comparison between randomization groups of patient safety, patient and endoscopist satisfaction, duration of patient recovery and of anesthesia procedure.

DETAILED DESCRIPTION:
What may be the benefits of general anaesthesia? In one retrospective study of more than 1000 patients, the ERCP failure rate with general anaesthesia was half compared to that observed with moderate sedation (7% versus 14%), with most failures resulting from inadequate sedation. It has also been reported that complication rates associated with therapeutic interventions during ERCP may be significantly lower when general anaesthesia is used, perhaps because the absence of patient movement makes the procedure technically less difficult. When general anaesthesia is administered for ERCP, the airway is protected by endotracheal intubation which may decrease risk for broncho-aspiration in some patients, although this measure has not been demonstrated to be effective in patients at risk during digestive endoscopy.

However, aspiration at the time of in/ex-tubation as well as micro-aspiration of contaminated upper airway secretions along leaks and defects of the tracheal cuff seal is not excluded if standard endotracheal tubes are used.

What may be the harms of general anaesthesia? Intubation and extubation manoeuvres may prolong endoscopic room occupation time, post-anaesthesia care unit stay may be longer and about 30 to 70% of patients will suffer from sore throat (this is reduced if lidocaine is used).

Furthermore, orotracheal intubation may induce short time hemodynamic changes related to laryngoscopy.

What may be the benefits of deep sedation? The main advantage of sedation is probably the faster turnover in the intervention room. In the sole practice survey of anesthesiologists for endoscopy that is available, 81% of anaesthesiologists stated that they were using sedation, not general anesthesia, for ERCP.

Deep sedation with propofol during digestive endoscopy has been shown to be superior to moderate sedation with a combination of benzodiazepine plus opioid in many aspects, including better patient cooperation, shorter recovery time and lower number of desaturation events.

In Switzerland, sedation during ERCP is obtained using benzodiazepines or propofol in similar proportions of cases and, when propofol is used, it is administered by the endoscopist or nurse in two thirds of cases and by the anaesthesiologist in one third of cases.

Evidence from prospective studies suggests that complex procedures, including therapeutic ERCP, may be performed safely under deep sedation without tracheal intubation using propofol, even in high-risk patients.

What may be harms of deep sedation? In a large study including nearly 10'000 patients, adverse events were observed in 1.4% of patients sedated using propofol. In that study, adverse events were defined as premature termination of the procedure due to sedation-related events (most often related to hypoxemia) or the need for assisted ventilation or, very rarely, admission to intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient with scheduled therapeutic ERCP
* Written informed consent for the study protocol obtained from the patient or his/her legal representative
* Anaesthetist available for the procedure

Exclusion Criteria:

* Mechanically ventilated patients before the procedure
* Baseline oxyhemoglobin saturation < 90%
* Baseline systolic blood pressure < 90 mm Hg
* American Society of Anaesthesiologists (ASA) physical score 5 (Table 1)
* Age < 18 years
* Pregnancy
* Emergency procedure
* Absence of fasting ≥ 6 hours for solids and ≥ 2 hours for clear liquids
* Contraindication to any study drug
* Short, thick neck or trismus that may complicate airway rescue
* Previous documented difficult airway intubation
* Obstructive sleep apnea
* Severe swallowing disorders with documented broncho-aspiration
* Bowel obstruction
* Inclusion in the present protocol during the 30 preceding days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-02; Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
ERCP success rate | 24 hours
  The primary study outcome will be a comparison between patient allocation groups and the percentage of completely successful ERCP. Success of ERCP is defined as achieving both high completion and low adverse event rate.

SECONDARY OUTCOMES:
Success of ERCP in subgroups of patients | 24 hours
  Secondary outcome will include a comparison between patient allocation groups of the success of ERCP in subgroups of patients (difficulty grade of ERCP = 2 or 3, ASA score = 4)

OTHER OUTCOMES:
composite "efficacy-safety" index | 30 days
  A composite "efficacy-safety" index will be calculated by adding the incidence, within 30 days of study ERCP, of repeat bilio-pancreatic procedure, major complication, re-hospitalisation and death.
patient satisfaction | 30 days
clinician satisfaction | 30 days
duration of patient recovery | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Huberty, MD, Principal Investigator — Gastroenterology Department Erasme Hospital
Locations (1):
- Gastroenterology Department Erasme Hospital, Brussels, Belgium